CLINICAL TRIAL: NCT00137748
Title: Does Replacement With CMVIG in Hypogammaglobulinemic Patients Decrease the Rate of Opportunistic Infections and Chronic Rejection?
Brief Title: Cytomegalovirus Hyperimmune Globulin (CMV-Ig) Replacement in Hypogammaglobulinemic Lung Transplant Recipients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB2953
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Hypogammaglobulinemia
Keywords: Lung transplantation
MeSH Terms: conditions — Agammaglobulinemia

INTERVENTIONS:
Drug: CMV-Ig — Drug: CMV-Ig

SUMMARY:
This is a randomized controlled trial of CMV-Ig in lung transplant recipients at the Cleveland Clinic Foundation who are hypogammaglobulinemic.

DETAILED DESCRIPTION:
This is a randomized controlled trial of CMV-Ig in lung transplant recipients at the Cleveland Clinic Foundation who are hypogammaglobulinemic.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant
* Hypogammaglobulinemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2001-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
CMV infection

CONTACTS AND LOCATIONS:
Overall Officials: Jeff T Chapman, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States